CLINICAL TRIAL: NCT05188157
Title: Mirror Therapy is an Adjuvant Treatment Option Based on Shoulder Impingement Syndrome.
Brief Title: Mirror Therapy for Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MLeblebicier2
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-12

CONDITIONS: Impingement Syndrome; Mirror Movements 2
Keywords: mirror therapy; Impingement Syndrome; shoulder; adjuvant treatment
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): conventional physiotherapy
  Interventions: Other: conventional physiotherapy
- mirror therapy group (Experimental): conventional physiotherapy and mirror therapy
  Interventions: Other: mirror therapy; Other: conventional physiotherapy

INTERVENTIONS:
Other: mirror therapy — The patients in IG will receive exercise program before mirror theraphy. The patient will continue to do the exercises in front of the mirror for the remaining 20 minutes of the exercise. While doing the exercise with the healthy side in front of the mirror, the patient will try to do the same movement with the shoulder diagnosed with impingement syndrome on the other side of the mirror. The patient will try to do the movement correctly with the reflection in the mirror.
  Arms: mirror therapy group
Other: conventional physiotherapy — The conventional physiotherapy program included, wand exercises for shoulder abduction, flexion, hyperextension and internal and external rotation, Codman exercises and isometric and resistive exercises of the shoulder girdle. The exercise program is performed under the supervision of an experienced physiotherapist. The isometric exercises will be used during the painful period, and the resistance exercises will be added after the pain began to relieve.under the supervision of a physician in the first 30 minutes of their exercise.

SUMMARY:
Background: Mirror therapy is an adjuvant treatment option based on shoulder impingement Syndrome Objective:To investigate the effect of mirror theraphy on shoulder impingement Syndrome Methods: The study included 62 participants, including cases in the intervention group (IG) (± years) and 20 cases in the control group (CG) (years) who met the selection criteria. IG received mirror theraphy with regular physiotherapy while CG received only regular physiotherapy. The patients were evaluated with the before treatment, immediately after treatment (post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18-75 years
* Being diagnosed with shoulder impingement syndrome

Exclusion Criteria:

* Being uncooperative
* Having an additional systemic disease
* Having uncontrolled hypertension
* Presence of heart failure
* Having hearing or vision problems
* Having a balance disorder
* Diagnosis of heart disease and lung disease so advanced that exercise is contraindicated
* History of shoulder surgery
* Have any pathology that may cause referred pain (eg, cervical radiculopathy)
* Shoulder trauma, previous humeral fracture history
* Steroid injection to the shoulder joint or subacromial bursa in the last 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
goniometer | 10 minutes
  shoulder range of motion and will be measured
Hawkins test | 5 minutes
  impingement tests; forced internal rotation was performed while the arm and elbow were in 90° flexion
Neer test | 5 minutes
  subacromial impingement test
Jobe Test | 5 minutes
  lesions of the infraspinatus muscle
Constant Murley Score | 10 minutes
  functional level of the patients' shoulder joint, higher scores mean a better outcome.
Tampa Kinesiophobia Scale | 10 minutes
  will be used to evaluate kinesiophobia, higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)